CLINICAL TRIAL: NCT07178743
Title: Emulation of the PALOMA-2 Trial
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor, Brigham and Women's Hospital
Other Study IDs: 2022P002556-ENC-PALOMA2; 75F40122C00181 (Other Grant/Funding Number: Food and Drug Administration)
Record Dates: First submitted 2025-09-08; First posted 2025-09-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-09

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Letrozole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Initiation of palbociclib plus letrozole: Exposure group
  Interventions: Drug: Initiation of palbociclib plus letrozole
- Initiation of letrozole: Reference group
  Interventions: Drug: Initiation of letrozole

INTERVENTIONS:
Drug: Initiation of palbociclib plus letrozole — Initiation of palbociclib plus letrozole described in electronic health records is used as the exposure.
  Groups: Initiation of palbociclib plus letrozole
Drug: Initiation of letrozole — Initiation of letrozole described in electronic health records is used as the reference.
  Groups: Initiation of letrozole

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale emulation of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
Randomized controlled trials (RCTs) are generally regarded as the gold-standard of evidence for establishing efficacy of medical products. However, real-world data (RWD) are increasingly used to complement evidence from RCTs. Yet, to have confidence in the accuracy of non-interventional studies medical products and their outcomes in oncology, investigators need to know what questions can be validly answered, with which non-interventional study designs, and which analysis methods are appropriate, given the data that is available. Building on a process from the RCT DUPLICATE initiative. EmulatioN of Comparative Oncology trials with Real-world Evidence (ENCORE) is the trial emulation discussed in this protocol is part of the expansion project specific to oncology and aims to emulate 12 randomized oncology RCTs using multiple EHR data sources.

The purpose of this protocol is to describe the emulation of the PALOMA-2 trial. PALOMA-2 was a Phase III, double-blind, randomized study assessing the efficacy and safety of palbociclib (125 mg orally, once daily for 21 days of a 28-day cycle) in combination with letrozole (2.5 mg orally, once daily, continuously) versus letrozole alone in postmenopausal women with estrogen receptor-positive (ER+), human epidermal growth factor receptor 2-negative (HER2-) advanced breast cancer who had not received prior systemic treatment for their advanced disease.

ELIGIBILITY:
Study Period:

ENCORE database 1 (EDB1): Patient identification period: 01/01/2011-04/30/2024 with follow-up information through data cut-off date on 04/30/2024

ENCORE database 3 (EDB3): Follow-up information through June 2023 (there is no specific time period restrictions for patient eligibility)

ENCORE database 4 (EDB4): Patient identification period: 10/01/2018-09/30/2023 with follow-up information through data cut-off date on 09/30/2023.

Inclusion Criteria:

* Age ≥18 years
* Postmenopausal women with ER-positive, HER2-negative locally advanced or metastatic breast cancer who receive treatment without curative intent
* The line of therapy for patients in EDB1 and EDB3 is implicitly advanced/metastatic because the line of therapy classification starts after their advanced/metastatic diagnosis in the respective database
* In EDB4, patients must explicitly have any evidence of a metastasis prior initiating palbociclib plus letrozole or letrozole alone
* Adenocarcinoma histology
* No prior systemic treatment for advanced/metastatic disease
* ECOG performance status of 0 or 1

Exclusion Criteria:

* HER2+
* CNS metastases
* Prior treatment with CDK4/6 inhibitor
* Non-breast cancer malignancy other than basal/squamous cell skin cancer or carcinoma in situ of cervix
* Systemic anticancer therapy other than palbocicilib or letrozole
* Treatment with non-steroidal aromatase inhibitor (i.e.anastrozole, letrozole)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with ER-positive, HER2-negative locally advanced or metastatic breast cancer who receive treatment without curative intent
Sampling Method: Non-Probability Sample
Enrollment: 6097 (Actual)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Time to all-cause mortality (overall survival) | Through the earliest of outcome, censoring, or end of data (April 2024)
  Hazard ratio (95% CI)

SECONDARY OUTCOMES:
Time to next treatment (TTNT) | Through the earliest of outcome, censoring, or end of data (April 2024)
  Median overall survival time (difference) in % (95% CI)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital; Denys Shay, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol (2025-08-18): https://cdn.clinicaltrials.gov/large-docs/43/NCT07178743/Prot_000.pdf